CLINICAL TRIAL: NCT00728910
Title: Combined Effects of Non-statin Treatments on Apolipoprotein A-I Up-Regulation (CENTAUR): A Feasibility Study
Acronym: CENTAUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Richard Dunbar, Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 807965 CNTR; CTRC #1123 (Other: University of Pennsylvania)
Record Dates: First submitted 2008-08-04; First posted 2008-08-06 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Dyslipidemia
Keywords: Low HDL cholesterol; High triglycerides; niacin; fibrate
MeSH Terms: conditions — Dyslipidemias; Hypertriglyceridemia | interventions — Atorvastatin; 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atorvastatin (Active Comparator): atorvastatin 10 mg/day by mouth for a total duration of 4 weeks
  Interventions: Drug: Atorvastatin
- ABT335 (Active Comparator): ABT335 135 mg/day by mouth added to atorvastatin for a total duration of at least 8
  Interventions: Drug: Atorvastatin; Drug: ABT335
- ER niacin (Active Comparator): ER niacin titrated up to 2 g/day with aspirin 325 mg/day by mouth added to atorvastatin and ABT335 for 10 weeks
  Interventions: Drug: Atorvastatin; Drug: ABT335; Drug: ER Niacin

INTERVENTIONS:
Drug: Atorvastatin — 10 mg QD for 4 weeks
  Other Names: Lipitor
Drug: ABT335 — 135 mg QD added to atorvastatin for 8 weeks
  Other Names: Trilipex
  Arms: ABT335; ER niacin
Drug: ER Niacin — 2000 mg QD added to atorvastatin and ABT335 for 10 weeks
  Other Names: Niaspan
  Arms: ER niacin

SUMMARY:
The investigators propose to investigate if using a combination of medications that may improve cholesterol give additional benefit to that gained from the statin medication, Lipitor. It is recommended that patients who meet certain criteria for risk of heart disease take a statin medication to improve cholesterol and hopefully reduce risk of heart disease. The combination therapy will include Lipitor, Niaspan, and investigational medication (known as ABT335) in a class of drugs called fibrates. We are looking to see if and how these three medications together might improve risk factors for atherosclerosis and influence HDL cholesterol. The study will also look at the safety and any side effects that might be associated with this combination of medications.

DETAILED DESCRIPTION:
Objectives Summary

* To investigate whether the progressive addition of a fibrate and niacin to baseline statin therapy will improve apolipoprotein A-I kinetics, postprandial lipidemia, and postabsorptive lipoproteins and metabolism in adult men and women with atherogenic dyslipidemia.

Major Efficacy Aims

* Objective 1 is to test the hypothesis that the fibrate ABT335 and extended release (ER) niacin progressively improve apolipoprotein A-I kinetics when added sequentially to baseline therapy with atorvastatin. The key outcomes include the apolipoprotein AI rate of catabolism and rate of production.
* Objective 2 is to test the hypothesis that the fibrate ABT335 and ER niacin progressively improve postprandial lipidemia by oral fat challenge when added sequentially to baseline therapy with atorvastatin. Key outcomes include the incremental area under the curve for triglycerides and high-density lipoprotein cholesterol.
* Objective 3 is to test the hypothesis that the fibrate ABT335 and ER niacin progressively improve markers of postabsorptive lipoproteins and metabolism when added sequentially to baseline therapy with atorvastatin. Key outcomes include a. fasting cholesterol efflux, b. HDL cholesterol, apolipoprotein A-I, and enzymes that remodel HDL, c. atherogenic lipoproteins, and d. markers of energy metabolism and e. markers of inflammation.

Additional Aims

* Objective 4 is to assess tolerability and adverse events when ABT335 and ER niacin are added sequentially to atorvastatin. Specifically, we will assess changes in hepatobiliary laboratory tests (including incidence of elevation), incidence of symptomatic myalgia, and incidence of flushing. On an exploratory basis, we will enhance the flushing evaluation with objective and subjective measurements of flushing during inpatient visits.

Study Design:

This is an open-label feasibility study of fixed-sequence addition of lipid-altering medications, in which comparisons are made to the baseline for each subject. Subjects begin a lead-in phase in which they start the study statin (atorvastatin) or switch from previous statin therapy to the study statin. Subjects will wash off other excluded lipid-altering drugs during the lead-in. Subjects return for the first inpatient visit, where they have baseline studies on statin monotherapy. At the end of this visit, subjects are started on fibrate therapy (ABT335). They repeat the studies on dual therapy with statin and fibrate, and then add niacin (ER niacin). To minimize flushing during chronic treatment, they start aspirin 325 mg daily, or titrate to 325 mg if they are taking a lower dose of aspirin (e.g. 81 mg). Finally, they repeat the studies on triple therapy with statin, fibrate, and niacin/aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. Men/women aged 18-80 years.
2. Low HDL-C, adjusted for baseline statin use

   1. Not on statin: Men with HDL <= 40 or women with HDL <= 50 mg/dL
   2. On statin: Men with HDL <= 42 or women with HDL <= 52 mg/dL
3. TG/HDL ratio >= 3.5
4. Able to understand and agree to informed consent
5. Women of child-bearing age must test negative on a urine pregnancy test and agree to use reliable birth control during the study and for 1 month after last dose of study drugs. Reliable methods include oral contraceptives, a barrier method, intrauterine device, partner with vasectomy, or abstinence.
6. Willing to be available for study duration and follow study procedures

Exclusion Criteria:

1. Subjects with following lipoprotein disorders:

   1. Patients on high-potency lipid-lowering regimen, defined as two or more prescription lipid-altering medications (excluding fish oils) where one is a high-dose statin (40 mg/day of rosuvastatin, 80 mg/day of other approved statins). Those on combination therapy with a lower statin dose or those taking high-dose statin monotherapy (excluding fish oils) may participate. Patients will switch to atorvastatin 10 mg and/or wash off other lipid medications to participate
   2. LDL > 190 mg/dL
   3. TG > 750 mg/dL or pancreatitis from triglyceridemia, regardless of current TG levels
   4. Dysbetalipoproteinemia (VLDL/TG > 0.3 -AND- TG > 200 mg/dL).
2. Use of non-statin lipid therapy prior to study initiation is exclusionary if (n.b. washout of non-statins is permitted):

   1. Niacin > 250 mg/ day within 6 weeks: Advicor, Niaspan, Niacor, Simcor, Slo-Niacin, or supplemental niacin
   2. Fibrates within 12 weeks: fenofibrate (Antara, Lofibra, Tricor, Triglide), gemfibrozil (Lopid), or clofibrate
   3. Enterically active drugs within 4 weeks: colestipol, cholestyramine, colesevelam, ezetimibe, orlistat.
   4. Red yeast rice during the treatment phase of the study (i.e. must be switched to study statin)
   5. Fish oil > 2 g/day within 4 weeks: Lovaza (née Omacor), numerous supplements
   6. Altered dose of a selective estrogen receptor modulator (SERM) within 4 weeks
3. Intolerance to statin, fibrate, aspirin, deuterated leucine, or niacin
4. Contraindications to medications, including chronic muscle disease, history of rhabdomyolysis, moderate-severe gout, severe peptic ulcer disease, bleeding disorders, and aspirin-sensitive asthma.
5. Diabetics, or fasting glucose > 110 mg/dL on two different days during screening, or use of anti-diabetic medications within 6 weeks of screening visit
6. Chronic renal insufficiency, nephrotic syndrome, or current serum creatinine > 2.5 mg/dL, or GFR < 60 mL/min/1.73m2 by the MDRD equation.
7. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin > 2 X the upper limit of normal (ULN), albumin of < 2.5 mg/dL, prothrombin time (PT) > 1.5 X ULN, partial thromboplastin time (PTT) > 1.5 X ULN, or current active hepatobiliary disease
8. Hemoglobin (Hgb) < 10 mg/dL
9. Weight < 110 lbs
10. Use of an investigational drug within 6 weeks prior to screening visit
11. Major surgery within the previous 6 weeks, or anticipated major surgery during course of study, or any history of organ transplant
12. Non-skin malignancy within previous 5 years
13. Drug abuse within past 3 years, or regular alcohol use >14 drinks/week
14. Women who are pregnant, plan to conceive, or breast-feed
15. Any serious or unstable medical or psychological conditions that, in investigator's opinion would compromise subject safety or successful participation.
16. Currently adhering to, planning to adhere to or used within 3 months prior to screening, supplements intended for weight loss or adopt diets with aggressive carbohydrate restrictions, such as but not limited to Atkins or South Beach diets.
17. Currently taking Vitamin A supplements (multivitamins allowed)(washout permitted)
18. Excluded concomitant medications

    1. Immunosuppressants within 2 months prior to screening or are likely to require such treatment during the course of the study
    2. Warfarin.
19. Disinclination to dairy products (e.g. inviolable dietary restrictions or lactose intolerance to an 8oz glass of milk despite lactase supplementation) Lactase supplementation is allowed during the study.
20. Regular consumers of grapefruit juice, or currently taking medications metabolized by CYP 3A4 (cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, and nefazodone)
21. History of pancreatitis or gallbladder disease
22. History of coronary heart disease
23. History of intolerance/adverse reaction to heparin or women who have dysfunctional uterine bleeding
24. Thrombocytopenia at screening
25. History of intracerebral or significant GI bleed
26. Subjects doing regular strenuous activity or have a CK > 3x ULN at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Dunbar, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- CTRC (Clinical Translational Research Center), Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted from June 2008 until February 2009.
Pre-assignment Details: Subjects washed out of current lipid lowering medications
Groups:
- Atorvastatin/ABT335/Niaspan: All participants received atorvastatin 10 mg/day for 4 weeks, followed by sequential addition of ABT335 135 mg/day for 8 weeks, and ER niacin 2000 mg/day for 10 weeks, for a total study duration of 22 weeks
Period: Atorvastatin
Arm/Group | Atorvastatin/ABT335/Niaspan
Started | 25
Completed | 22
Not Completed | 3
Period: Atorvastatin+ABT335
Arm/Group | Atorvastatin/ABT335/Niaspan
Started | 22
Completed | 22
Not Completed | 0
Period: Atorvastatin+ABT335+ER Niacin
Arm/Group | Atorvastatin/ABT335/Niaspan
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: All participants received atorvastatin 10 mg/day for 4 weeks, followed by sequential addition of ABT335 135 mg/day for 8 weeks, and ER niacin 2000 mg/day for 10 weeks.
Arm/Group | Group 1
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Apolipoprotein A-I Fractional Catabolic Rate (FCR)
Description: After receiving total daily caloric intake over 20 hrs as 20 identical small meals, starting at 0600 hrs, subjects took study medications at 0800 hrs. Five hours after the first meal, i.v. 5,5,5-2H3-L-leucine was administered, followed by a primed-constant infusion at 10 mol/kg body weight per hr for 15 hrs during which 14 blood samples were collected. Isotopic enrichment of leucine in apoA1 band excised from polyacrylamide gel was calculated. Assuming steady state apo A-I metabolism, we used a compartment model to fit data, consisting a precursor compartment (Compartment 1), the plasma leucine pool, an intracellular compartment accounting for apoA1 synthesis and lipoprotein assembly (Compartment 2), and compartments to account for dispositional kinetics of the subfractions including a plasma pool compartment (Compartment 3). The apoA1 FCR corresponds to the rate of irreversible loss of leucine pools from Compartment 3.
Time Frame: 4 weeks, 12 weeks and 22 weeks
Population: Patients who completed any of the three phases for whom the kinetic study data was available for any phase of treatment
Measure: Mean (95% Confidence Interval); unit: pools/day
Groups:
- Atorvastatin: Subjects received atorvastatin 10 mg daily by mouth for 4 weeks followed by apo-A1 kinetics
- Atorvastatin+ABT335: Subjects received atorvastatin 10 mg daily and ABT335 135 mg daily by mouth for 8 weeks.
- Atorvastatin+ABT335+Niaspan: Subjects received atorvastatin 10 mg daily, ABT335 135 mg and Niaspan 2000 mg daily by mouth for 10 weeks.
Arm/Group | Atorvastatin | Atorvastatin+ABT335 | Atorvastatin+ABT335+Niaspan
Number analyzed (Participants) | 21 | 21 | 20
pools/day | 0.294 [0.27 to 0.32] | 0.294 [0.27 to 0.32] | 0.295 [0.25 to 0.34]
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+ABT335 vs Atorvastatin+ABT335+Niaspan; Null hypothesis was that the sequential addition of a fibrate and niacin to baseline atorvastatin therapy would not have any effect on apo-AI catabolism; Test type: Superiority or Other; p > 0.5, Mixed Models Analysis

2. Primary Outcome: Apo-A1 Production Rate
Description: The apolipoprotein A-I production rate using (5,5,5-2H3-L-leucine) was measured following each of the three study periods i.e following 4 weeks of atorvastatin 10 mg/day, following 8 further weeks of ABT335 135 mg/day added to atorvastatin and following 10 further weeks of ER niacin 2000 mg/day and aspirin 325 mg/day added to atorvastatin+ABT335.
Time Frame: 4 weeks, 12 weeks and 22 weeks
Population: Patients who completed any phase of treatment for whom kinetic data were available
Measure: Mean (95% Confidence Interval); unit: mg/kg/day
Arm/Group | Atorvastatin | Atorvastatin+ABT335 | Atorvastatin+ABT335+Niaspan
Number analyzed (Participants) | 20 | 20 | 20
mg/kg/day | 14.2 [11 to 17] | 14.2 [12 to 17] | 13.8 [11 to 17]
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+ABT335 vs Atorvastatin+ABT335+Niaspan; The null hypothesis was that sequential addition of fibrate and niacin to baseline atorvastatin therapy would have no effect on apo-A1 production rates; Test type: Superiority or Other; p > 0.5, Mixed Models Analysis

3. Primary Outcome: Post-prandial Triglyceride Incremental Area Under the Curve (iAUC)
Description: Triglyceride iAUC was measured during an oral fat tolerance test administered after 4 weeks of atorvastatin 10 mg/day , a further 8 weeks of atorvastatin 10mg /day+ABT335 135mg/day and then after a further 10 weeks of atorvastatin 10 mg/day+ABT335 135 mg/day+Niaspan 2000 mg/day. The standardized oral fat load was administered one hour post medication dosing and blood was collected prior to drug dosing, prior to the oral fat load and hourly thereafter for 10 hours (0,1,2,3,4,5,6,7,8,9,10,12 hrs post drug dosing)
Time Frame: 4 weeks, 12 weeks, 22 weeks
Population: subjects completing any phase of treatment for whom complete post-prandial data were available
Measure: Mean (95% Confidence Interval); unit: mg/dl*h
Groups:
- Atorvastatin: Subjects received atorvastatin 10 mg daily by mouth for 4 weeks followed by an oral fat tolerance test
- Atorvastatin+ABT335: Subjects received atorvastatin 10 mg daily and ABT335 135 mg daily by mouth for 8 weeks followed by an oral fat tolerance test.
- Atorvastatin+ABT335+Niaspan: Subjects received atorvastatin 10 mg daily, ABT335 135 mg and Niaspan 2000 mg daily by mouth for 10 weeks followed by an oral fat tolerance test.
Arm/Group | Atorvastatin | Atorvastatin+ABT335 | Atorvastatin+ABT335+Niaspan
Number analyzed (Participants) | 22 | 22 | 22
mg/dl*h | 770 [618 to 921] | 515 [361 to 670] | 381 [214 to 547]
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+ABT335; Null hypothesis was that sequential addition of fibrate and niacin to baseline atorvastatin therapy would have no effect on post-prandial triglyceride levels following an oral fat load; Test type: Superiority or Other; p < 0.0005, Mixed Models Analysis
Statistical Analysis 2: Comparison: Atorvastatin vs Atorvastatin+ABT335 vs Atorvastatin+ABT335+Niaspan; Test type: Superiority or Other; p < 0.0005, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 22 weeks
Groups:
- Atorvastatin/ABT335/Niaspan: Subjects received atorvastatin 10 mg/day for 4 weeks, followed by addition of ABT335 135 mg/day for a further 8 weeks followed by the addition of Niaspan 2000 mg/day for a further 10 weeks.
Arm/Group | Atorvastatin/ABT335/Niaspan
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin/ABT335/Niaspan (N=25)
ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin/ABT335/Niaspan (N=25)
headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No